CLINICAL TRIAL: NCT00638079
Title: Single-center, Randomized, Open-label, 2-way Crossover Bioavailability Study, Evaluating the Effect of Food on Megace ES (Megestrol Acetate 625 mg/5 mL Oral Suspension) Following a 625 mg Dose in Healthy Subjects
Brief Title: Evaluating the Effect of Food on Absorption of Megace ES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: SFBC Anapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PAR 100.1.C.003
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics; Bioavailability; Absorption
Keywords: Pharmacokinetics; Food Effect; Bioavailability; Megace ES
MeSH Terms: interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Megestrol acetate 625 mg/5 mL oral suspension (Megace ES) with a high fat meal
  Interventions: Drug: Megestrol acetate oral suspension 625 mg/5 mL
- B (Active Comparator): Megestrol acetate 625 mg/5 mL oral suspension (Megace ES) following an overnight fast
  Interventions: Drug: Megestrol acetate oral suspension 625 mg/5 mL

INTERVENTIONS:
Drug: Megestrol acetate oral suspension 625 mg/5 mL — Megestrol acetate oral suspension 625 mg/5 mL. Single dose (5 mL) administered with a high fat meal
  Other Names: Megace ES
  Arms: A
Drug: Megestrol acetate oral suspension 625 mg/5 mL — Megestrol acetate oral suspension 625 mg/5 mL. Single dose (5 mL) administered following an overnight fast
  Other Names: Megace ES
  Arms: B

SUMMARY:
To evaluate the effect of food on the rate and extent of absorption of megestrol acetate 625 mg/5 mL , and determine the safety and tolerability of megestrol acetate 625 mg/5 mL in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ranging from 60-100 kg (132-220 lbs) and body mass index ≥18 and ≤32
* Healthy

Exclusion Criteria:

* History of or any current medical conditions that could interfere with drug consumption, absorption, distribution, metabolism (eg. CYP450 inducers or inhibitors), or excretion of study drug
* History of or any current medical conditions that could affect subject safety
* History of frequent nausea or emesis, regardless of etiology
* Participation in a clinical drug study during the 30 days preceding the initial dose
* Significant illness during the 4 weeks preceding study entry
* Use of any medication, including vitamins/herbal/mineral supplements, during the 7 days preceding the initial dose
* Refusal or inability to abstain from food 10 hours proceeding and 4 hours following study drug administration, to consume the FDA high fat meal as directed, and to abstain from caffeine- or xanthine-containing beverages entirely during each confinement
* Any history of or current drug or alcohol abuse
* Prior alcohol intake exceeding the equivalent of 14 units/week (12 oz beer = 4 oz wine = 1.5 oz shot = 1 unit) on average, or consumption of any alcoholic beverages within 48 hours of study drug administration
* History of smoking>25 cigarettes/day within 45 days of study drug administration
* Blood or blood products donated within 30 days prior to study drug administration, or anytime during the study, except as required by this protocol
* Positive results of urine drug screen, blood alcohol by a Breathalyzer test, hepatitis B surface antigen, hepatitis B surface antibody (unless immunized), or anti-HCV

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 120 hours (5 days)
Safety assessed using adverse events (AEs), clinical laboratory results, vital signs, physical examinations, and ECGs. | signing of informed consent to 30 days after last study visit

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Deschamps, MD, Principal Investigator — SFBC Anapharm; Todd Kirby, PhD, Study Director — Endo Pharmaceuticals
Locations (1):
- SFBC Anapharm, Montreal (Quebec), Canada

REFERENCES:
- [Result] Deschamps B, Musaji N, Gillespie JA. Food effect on the bioavailability of two distinct formulations of megestrol acetate oral suspension. Int J Nanomedicine. 2009;4:185-92. doi: 10.2147/ijn.s6308. Epub 2009 Sep 10. PMID 19774117
- See also: International Journal of Nanomedicine — http://www.dovepress.com/international-journal-of-nanomedicine-journal